CLINICAL TRIAL: NCT02832206
Title: EndoMaze HYBRID project-a Detailed Assessment of Efficacy and Safety of Hybrid Ablation of Persistent and Long-standing Persistent Atrial Fibrillation
Brief Title: Hybrid Ablation of Persistent and Long-standing Persistent Stand-alone Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Petr Budera, M.D., Ph.D., Charles University, Czech Republic
Other Study IDs: PRAGUE-21
Record Dates: First submitted 2016-06-29; First posted 2016-07-14 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Hybrid ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- hybrid ablation: 60 patients with stand-alone, persistent or long-standing persistent atrial fibrillation
  Interventions: Procedure: hybrid ablation

INTERVENTIONS:
Procedure: hybrid ablation — Surgical thoracoscopic epicardial ablation (box-lesion) and left atrial appendage occlusion , followed (after 2-3months) by electrophysiological examination, and catheter ablation (completion of the box-lesion, cavotricuspid isthmus ablation and other ablation if indicated)

SUMMARY:
This study evaluates in detail efficacy and safety (including neurological safety) of hybrid ablation of stand-alone, persistent and long-standing persistent atrial fibrillation (AF). An implantable ECG monitor will be implanted to all patients for rhythm monitoring. Neurological safety will be assessed by cerebral magnetic resonance, neuropsychological examination and periprocedural transcranial Doppler measurement.

DETAILED DESCRIPTION:
Hybrid ablation (i.e. surgical thoracoscopic ablation, followed by catheter endocardial ablation) represent a new treatment option for patients with atrial fibrillation.

60 patients will undergo a two-stage, hybrid ablation, all of them will have an ECG monitoring device implanted and will be followed for up to three years. Neurological safety of both surgical and catheter procedures will be assessed by three examinations. Magnetic resonance will be performed before surgery, 5 days after surgery and at the 180 days visit to search for (subclinical) cerebral ischemia. Complex neuropsychological examination will be performed before surgery, afer 1 month after surgery and at 180 days visit to search for changes in cognitive functions, behavioral functions etc. Transcranial Doppler will be performed during surgical and catheter ablation to detect microembolic signals.

ELIGIBILITY:
Inclusion Criteria:

* Patients age > 18 years
* Patients with persistent/long-standing persistent AF according to the standard EHRA definition.
* Patients with symptomatic AF that is refractory to at least one antiarrhythmic medication.
* Absence of significant structural heart disease (dilated cardiomyopathy, hypertrophic cardiomyopathy, valvular heart disease, untreated coronary artery disease)
* Ability to sign an informed consent

Exclusion Criteria:

* Paroxysmal AF
* AF secondary to a reversible cause (i.e., thyreopathy, etc.)
* Indication for open-heart surgery (coronary artery bypass grafting, valve surgery, etc.)
* Severe left ventricle dysfunction that is clearly caused by some other cardiac disease (dilated cardiomyopathy, ischaemic heart disease, etc.) where the AF is clearly of secondary etiology
* Known severe pericardial and pleural adhesions (e.g., history of cardiac surgery)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with symptomatic, drug-resistant, stand-alone, persistent or long-standing persistent atrial fibrillation
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
sinus rhythm (The Reveal LINQ Insertable Cardiac Monitoring System) | 1 year
  Number of patients with sinus rhythm, without detections of atrial arrhythmias (episodes longer than 30 seconds)

SECONDARY OUTCOMES:
neurological safety (cerebral magnetic resonance (MR), neuropsychological changes - multiple questionnaires, Transcranial Doppler) | 180 days
  new ischaemic brain lesions on MR performed at the discharge from surgery and at the 180 days visit), neuropsychological changes measured by special questionnaires, that will be filled at 30 and 180 days visit, periprocedural Doppler - hits rates on periprocedural transcranial Doppler measurement during both surgery and catheter ablation
periprocedural complications - surgery | 30 days
  conversion to sternotomy, bleeding, thromboembolic events, tamponade, haemothorax, pneumothorax, pleural effusion, pneumonia

OTHER OUTCOMES:
QoL measurement | 1 year
  changes in quality of life, measured by questionnaires AFEQT

CONTACTS AND LOCATIONS:
Overall Officials: Zbynek Straka, MD, PhD, Principal Investigator — University Hospital Kralovske Vinohrady
Locations (1):
- Charles University, Third Faculty of Medicine, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Osmancik P, Budera P, Zdarska J, Herman D, Petr R, Fojt R, Straka Z. Residual echocardiographic and computed tomography findings after thoracoscopic occlusion of the left atrial appendage using the AtriClip PRO device. Interact Cardiovasc Thorac Surg. 2018 Jun 1;26(6):919-925. doi: 10.1093/icvts/ivx427. PMID 29360987